CLINICAL TRIAL: NCT01787578
Title: A Prospective Safety, Tolerance, Pharmacodynamics and Pharmacokinetics Study of Sobetirome in Male Subjects Diagnosed With X-linked Adrenoleukodystrophy (X-ALD)
Brief Title: Safety and Pharmacodynamic Study of Sobetirome in X-Linked Adrenoleukodystrophy (X-ALD)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: revisions to original study protocol underway
Sponsor: Thomas S. Scanlan (Other)
Responsible Party: Sponsor-Investigator, Thomas S. Scanlan, Professor of Physiology & Pharmacology, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobetirome-CLIN-006; CTSA grant (UL1TR000128) (Other Grant/Funding Number: Oregon Clinical & Translational Research Institute)
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: X-Linked Adrenoleukodystrophy; Adrenomyeloneuropathy
Keywords: X-linked adrenoleukodystrophy; adrenomyeloneuropathy; sobetirome; thyroid; thyromimetic
MeSH Terms: conditions — Adrenoleukodystrophy; Thyroid Diseases | interventions — GC 1 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sobetirome (Experimental): Subjects will receive oral doses of sobetirome. All subjects will start with a 50 mcg dose, once-daily for 14 days. If this dose proves safe and well tolerated, subjects will receive a 100 mcg dose once-daily for an additional 14 days.
  Interventions: Drug: Sobetirome

INTERVENTIONS:
Drug: Sobetirome — 50 mcg or 100 mcg once-daily oral
  Other Names: GC-1; QRX-431

SUMMARY:
The purpose of this study is to assess the safety, tolerance, pharmacokinetics, and pharmacodynamics of sobetirome, a selective thyroid hormone analog, in adult male X-ALD patients.

DETAILED DESCRIPTION:
Subjects will have a screening visit within 6 weeks prior to the Baseline visit. At Baseline visit blood will be drawn and to establish baseline values for plasma and red blood cell (RBC) very long chain fatty acids (VLCFA; C22, C24, and C26). Subjects will receive an oral dose of 50 mcg sobetirome once daily for 14 days beginning on Day 1. Subjects will be kept in the clinic on Day 1 for 16 hours following their initial dose of sobetirome for repeat blood sampling for pharmacokinetic analysis. Subjects will return to the clinic on days 7, 15, 21 and 28 for blood collection for VLCFA measurements. On day 15, after safety assessment, subjects will receive an increased dose of 100 mcg and this dose will be continued once daily through Day 28. Subjects will continue to return to the clinic weekly for blood and urine collection and safety assessments. Subjects will return to the clinic on day 42 for an End of Study visit that will involve a final measurement of VLCFA and blood and urine safety labs to check for reversibility. Safety labs will include serum chemistry, free fatty acid profile, hematology, urinalysis, and thyroid function. Subjects will be monitored with ECGs, vital signs, physical exams and assessment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* males 18-65 years old
* X-ALD diagnosis by either elevated VLCFAs or DNA testing
* must sign informed consent and agree to complete required clinic visits.

Exclusion Criteria:

* female gender
* abnormal laboratory test results (except VLCFA) at screening visit
* history of coronary artery disease
* use of triiodothyronine therapy
* abnormal thyroid function test at screening visit
* untreated adrenal insufficiency
* currently taking Lorenzo's Oil or other VLCFA lowering agent
* participation in investigational drug study within 30 days

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Estimated); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in very long chain fatty acid (VLCFA) levels | Day 14 and Day 28 of sobetirome dosing
  Very long chain fatty acid (VLCFA) levels in plasma and erythrocytes will be measured after 14 days of 50 mcg sobetirome, and again after 14 days of 100 mcg sobetirome dosing.

SECONDARY OUTCOMES:
Evidence of changes in thyroid function from baseline confirmed by measured changes in TSH and/or free T4 | Day 14 and 28 of sobetirome dosing
  Thyroid function will be assessed my measurement of TSH and free T4 following 14 days of 50 mcg sobetirome, and again following 14 days of 100 mcg sobetirome dosing.
Number of participants with adverse events from baseline | Every 7 days to outcome visit day and again at end of study visit day
  Adverse events will be assessed by physical examination and ECG
Peak Plasma Concentration (Cmax) of Sobetirome | Day 1
  A pharmacokinetic analysis to assess sobetirome exposure in X-ALD subjects.

CONTACTS AND LOCATIONS:
Overall Officials: David Koeller, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States